CLINICAL TRIAL: NCT03285867
Title: Value of Liver Stiffness Measurement (LSM) in Predicting the Progress of Liver Fibrosis After Transcatheter Arterial Chemoembolization (TACE) for Hepatocellular Carcinoma, an Observational Study
Brief Title: Liver Stiffness Measurement (LSM) in Predicting Progress of Liver Fibrosis After TACE for Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: liuhy
Record Dates: First submitted 2017-08-27; First posted 2017-09-18 (Actual); Last update posted 2018-04-30 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma; Liver Failure
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HCC received TACE: observational study set only one group with HCC received TACE
  Interventions: Procedure: TACE

INTERVENTIONS:
Procedure: TACE — transcatheter arterial chemoembolization

SUMMARY:
Objective: To evaluate the efficacy of preoperative liver stiffness measurement(LSM) by FibroScan in predicting the progress of liver fibrosis and prognosis after transcatheter arterial chemoembolization (TACE) in hepatocellular carcinoma (HCC).

Background: Progress of liver fibrosis and liver failure and related poor prognosis after TACE which are not completely predictable by current method including Child-Pugh Classification. LSM is used to calculate the degree of liver fibrosis and is affected by several liver injury, e.g. elevated Alanine aminotransferase（ALT）, Aspartate transaminase(AST) and Bilirubin et al. The investigators assume that LSM could be use to predict progress of liver fibrosis and adverse effects after TACE in HCC.

Methods: At least 200 patients will be recruited in this prospective observational study with preoperative LSM, demographic, laboratory, radiological and other treatment-related factors. Participants will be followed up till death or to the end of study no matter the liver failure occurs or not. Data will be analyzed to build a mathematical predicting model.

Research hypothesis：TACE is related to progress of liver fibrosis and a mathematical model with LSM is able to predict the risk of liver failure and prognosis in HCC.

ELIGIBILITY:
Inclusion Criteria:

* age：18-80
* HCC diagnosed by pathologist or physician according to Guidelines
* Chronic Hepatitis B (CHB) background
* receive at least 1 TACE
* volunteer to join the research

Exclusion Criteria:

* massive lesion with insufficient liver left for LSM examination
* associated with other liver diseases: Chronic Hepatitis C(CHC),Autoimmune Hepatitis(AIH),Wilson's disease.
* severe obesity(BMI>28)
* pregnancy
* other inappropriate situation defined by investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients admitted to our department
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-06-25 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
The change of LSM(kpa) measured by FibroScan(a kind of external harmless ultrasonoscope) | within 1 week pre-TACE and 1 week post-TACE
  The investigators will investigate the value of LSM( kpa) by machine of FibroScan ( produced by France Echo).
  The investigators will record LSMs before and after each procedure of TACE. The investigators will calculate the change of LSMs of each participants.

IPD SHARING:
Plan to Share IPD: No